CLINICAL TRIAL: NCT04432935
Title: Effect of Bovine Lactoferrin on Seroconversion Following Polio Vaccine Administration in Children: A Randomized Control Trial
Brief Title: Effect of Lactoferrin on Polio Seroconversion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-1955-5013
Record Dates: First submitted 2019-12-11; First posted 2020-06-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Poliomyelitis
Keywords: Bovine Lactoferrin; Poliovirus; Routine immunization
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: Group 1:
  Bovine lactoferrin (bLF) will be administered (300mg) from day 0 of birth to 6 weeks of life with a single daily dose mixed with milk (preferentially breast milk otherwise premature formula milk).
  Group 2:
  Placebo will be administered from day 0 of birth to 6 weeks of life. (Placebo will be physically identical to the bLF mixed with breast milk or premature formula milk).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be carried out by Data management unit and all investigators /dispensers and participants will be masked to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bovine Lactoferrin (Experimental): Intervention group will receive bovine lactoferrin supplementation daily once a day from day 0 of birth to 6 weeks of life.
  Interventions: Dietary Supplement: Bovine Lactoferrin
- Glucon D (Placebo Comparator): Control group will receive Glucon-D supplementation daily once a day from day 0 of birth to 6 weeks of life.
  Interventions: Other: Placebo Glucon D

INTERVENTIONS:
Dietary Supplement: Bovine Lactoferrin — Lactoferrin is a nutritional supplement which was first discovered in bovine milk which was later isolated in human milk as the second most abundant protein; with high levels found in colostrum. The use of bovine Lactoferrin in children is generally recognized as safe by the US Food and Drug Administration.
  Arms: Bovine Lactoferrin
Other: Placebo Glucon D — This group will be given 100mg Glucon-D (99.4% glucose) which will be similar in shape, color to the bLF.
  Arms: Glucon D

SUMMARY:
A massive decline in cases of poliomyelitis was observed worldwide since 1988; however its transmission continues in Pakistan and Afghanistan. In 2017, a total of 17 cases were reported from these countries, which represent approximately half of the cases reported in 2016. This achievement was made possible by large scale use of oral polio vaccine (OPV) and inactivated polio vaccine (IPV). Despite vigorous efforts to end poliovirus transmission in endemic areas, several challenges including illiteracy, poverty, malnutrition, difficulty to access health and immunization services adversely affect the effectiveness of the polio eradication efforts. Innovations are thus needed to accomplish the goal of eradication as due to limited funding, the sustainability of a program becomes questionable. The aim of this study is to assess the effectiveness of lactoferrin in increasing mucosal and serum immunity in children following administration of poliovirus vaccines.

DETAILED DESCRIPTION:
Lactoferrin was first discovered in bovine milk which was later isolated in human milk as the second most abundant protein; with high levels found in colostrum. Evidence suggests that Lactoferrin enhances a child's immunity against gastrointestinal infections by inhibiting the growth of bacteria through iron deprivation and by preventing attachment of the virus to the intestinal cells thus children become less susceptible to virus replication in the gut. Investigations of enhanced efficacy of the BCG (Bacillus Calmette-Guérin) vaccine after administration of Lactoferrin showed promising results. The use of bovine Lactoferrin in children is generally recognized as safe by the US Food and Drug Administration. Its anti-infective properties creates a new window of opportunity to assess its effects on the level of seroconversion following poliovirus vaccination in children.

This is a double-blinded two arm randomized placebo-controlled trial. A total of 377 neonates will be enrolled in each group (754 neonates in both groups). Females ages 18-45 years in their last trimester of pregnancy in Karachi, Pakistan will be recruited for the study by the study team and consent will be obtained. Participants will be newborns (on day 1 of birth) who will be followed through 6 months of age. Newborns who fulfill the inclusion criteria will be randomly assigned to the control or intervention group in 1:1 ratio on the first day of birth. Intervention group will receive a daily bovine lactoferrin supplementation whereas Control group will receive a daily placebo supplementation along with breast milk from day 0 of birth to 6 weeks of life. Newborns will be followed up daily during the course of the hospital stay.

After discharge from the hospital, mothers will be provided with a week's supply of lactoferrin or placebo along with instructions on how and when to administer it to the baby. Newborns will be followed up weekly. Compliance will be assessed by counting the used sachets of lactoferrin or placebo because mothers will be instructed to keep the empty sachets in a dedicated container issued by study staff. Mothers will be strictly advised to administer all vaccinations according to the routine immunization schedule. For both groups, a blood sample will be collected in the hospital and containers will be given to the mother for collections of stool for the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females aged 18 to 45 years with no underlying complications or co-morbidities
* Residence less than 30 kms away from the study clinic and have resided there for at least 1 year. Family MUST indicate that they will not move from their current residence for the 5 months after birth of the child (study period)
* Healthy singleton full-term births born to these mothers, regardless of birth weight and an APGAR score of 7 or higher 5 minutes after delivery with no underlying complication (randomization will take place at this stage)

Exclusion Criteria:

* Females with health issues and high risk pregnancies
* Neonates presenting with any morbidities and congenital anomalies will be excluded from the study
* Preterm birth (<37 weeks of gestation)
* Immunodeficiency disorder in immediate family member
* Parents refusing to consent

Ages: 1 Hour to 23 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 468 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of humoral immunity by seroconversion | 10 weeks
  Presence of detectable antibodies to poliovirus types 1 and 3 in serum) after receipt of two doses of OPV

SECONDARY OUTCOMES:
Comparison of humoral immunity represented by seroconversion | 18 weeks
  Presence of detectable antibodies to poliovirus types 1, 2 and 3 in serum) after completion of the routine immunization doses/schedule
Comparison of intestinal immunity represented by shedding of poliovirus types 1 and 3 | 19 weeks
  If lactoferrin is effective in improving intestinal immunity, shedding is expected to be lower in the lactoferrin receiving group.
Comparison of duration of shedding among the two study arms | 20 and 22 weeks
  Represented by shedding at 20 weeks of age and at 22 weeks of age after the challenge dose of bOPV administered

CONTACTS AND LOCATIONS:
Overall Officials: Sajid Soofi, MBBS, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Kharadar Campus, Aga Khan University Hospital, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Study findings will be disseminated through presentations at scientific conferences and educational practice workshops and will be published in an international peer-reviewed scientific journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the manuscript has been prepared and published.
Access Criteria: A formal application to the PI will be required requesting him about the accessibility of the data. This should include the rationale and expected use of the study data.

REFERENCES:
- [Background] Hussain SF, Boyle P, Patel P, Sullivan R. Eradicating polio in Pakistan: an analysis of the challenges and solutions to this security and health issue. Global Health. 2016 Oct 12;12(1):63. doi: 10.1186/s12992-016-0195-3. PMID 27729081
- [Background] Roseanu A, Brock JH. What are the structure and the biological function of lactoferrin in human breast milk? IUBMB Life. 2006 Apr;58(4):235-7. doi: 10.1080/15216540600577897. No abstract available. PMID 16754302
- [Background] Seganti L, Di Biase AM, Marchetti M, Pietrantoni A, Tinari A, Superti F. Antiviral activity of lactoferrin towards naked viruses. Biometals. 2004 Jun;17(3):295-9. doi: 10.1023/b:biom.0000027708.27142.bc. PMID 15222481
- [Background] Ochoa TJ, Cleary TG. Effect of lactoferrin on enteric pathogens. Biochimie. 2009 Jan;91(1):30-4. doi: 10.1016/j.biochi.2008.04.006. Epub 2008 Apr 18. PMID 18472012
- [Background] Superti F, Ammendolia MG, Valenti P, Seganti L. Antirotaviral activity of milk proteins: lactoferrin prevents rotavirus infection in the enterocyte-like cell line HT-29. Med Microbiol Immunol. 1997 Oct;186(2-3):83-91. doi: 10.1007/s004300050049. PMID 9403835
- [Background] Hwang SA, Wilk KM, Budnicka M, Olsen M, Bangale YA, Hunter RL, Kruzel ML, Actor JK. Lactoferrin enhanced efficacy of the BCG vaccine to generate host protective responses against challenge with virulent Mycobacterium tuberculosis. Vaccine. 2007 Sep 17;25(37-38):6730-43. doi: 10.1016/j.vaccine.2007.07.005. Epub 2007 Jul 27. PMID 17698261
- [Background] Hwang SA, Arora R, Kruzel ML, Actor JK. Lactoferrin enhances efficacy of the BCG vaccine: comparison between two inbred mice strains (C57BL/6 and BALB/c). Tuberculosis (Edinb). 2009 Dec;89 Suppl 1:S49-54. doi: 10.1016/S1472-9792(09)70012-5. PMID 20006305
- [Derived] Habib A, Nausheen S, Nooruddin S, Javed T, Samejo T, Hussain A, Namdev S, Amirali S, Umer M, Sheikh L, Hussain I, Ariff S, Soofi S. Effect of bovine lactoferrin on seroconversion following polio vaccine administration in children: protocol for a double-blinded randomised controlled trial. BMJ Open. 2022 May 24;12(5):e050849. doi: 10.1136/bmjopen-2021-050849. PMID 35613782
- See also: Agency Response Letter GRAS Notice No. GRN 000611 — https://www.fda.gov/food/gras-notice-inventory/agency-response-letter-gras-notice-no-grn-000611